CLINICAL TRIAL: NCT04993326
Title: Advancing DSME/S and COVID-19 Prevention and Protection Through "emPOWERed to Change" Program
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not funded
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 1774297-1
Record Dates: First submitted 2021-08-04; First posted 2021-08-06 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Type2 Diabetes; Covid19
Keywords: Diabetes Education, African Americans, COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): emPOWERed to Change
  Online Courses:
  4 Critical Step to Manage Diabetes modules
  * Step 1 Learn about diabetes
  * Step 2 Know your diabetes ABCs
  * Step 3 Learn how to live with diabetes
  * Step 4 Get routine care to stay healthy Diabetes + COVID-19 Protection and Prevention modules
  * Introduction to understanding COVID-19 and the risks specific to T2DM
  * Learn preventive and protective measures to avoid COVID-19
  * COVID-19 Vaccine education and Discussion guide
  * Community resource guide to access COVID-19 testing and vaccination Stress Management modules
  * Understanding of the relationship between diabetes and stress
  * Learn stress management techniques for diabetes Ongoing Program Support: Motivation for participation, medication adherence, accountability and peer-to-peer interaction and support (bi-weekly text messages & private and closed Facebook community support group with peers and professionals)
  Interventions: Behavioral: emPOWERed To Change Program
- Control (No Intervention): Usual Standard of Care as deemed by participants provider(s)

INTERVENTIONS:
Behavioral: emPOWERed To Change Program — Online Diabetes Self-Management Education and Support along with COVID-19 prevention and protection (vaccination) education and resource information
  Arms: Intervention

SUMMARY:
African Americans (AA)/People of Color (POC) are disproportionately impacted by COVID-19 to an extent not observed in other racial/ethnic subgroups. People of color are uniquely affected because keeping diabetes under control - the best defense against COVID-19 - has become more difficult as the pandemic has disrupted medical care, exercise and healthy eating routines which are already well-known challenges for the African American community. Diabetes Self-Management Education and Support (DSMS/S) facilitates the knowledge, skills, and ability necessary for diabetes self-care as well as activities that assist a person in implementing and sustaining the behaviors needed to manage their condition on an ongoing basis. Now, given the implications of COVID-19 on the AA/POC diabetes community, it is imperative to enhance DSME/S with education about protection and prevention of COVID-19. To begin to solve this problem we will adapt and implement the "emPOWERed to Change" DSME/S program to provide enhanced type 2 diabetes mellitus (T2DM) education with an additional emphasis on COVID-19 protection and prevention. This study will employ Community Based Participatory Research methods and will be conducted virtually in the community setting. The proposed hypothesis, based on the Health Belief Model (HBM) and the Theory of Planned Behavior (TPB), is: African Americans (AA)/People of Color (POC) in Los Angeles County with type 2 diabetes mellitus (T2DM) randomized to participate in the "emPOWERed to Change" program (N=48) are more likely to demonstrate sustained glycemic control, increase in knowledge and skills related behaviors, and risk factors associated with T2DM and SARS-CoV-2 (COVID-19) and increased compliance with prevention, and vaccination as compared to those who are randomized to usual care (N=48) in this 12 week program. We propose a randomized control study design among 96 participants with 48 assigned to an intervention group and 48 assigned to a control group. This study will also explore the experience of the participants' appraisal of knowledge and skills acquisition for DSME/S to maintain T2DM control, reduce complications, and SARS-CoV-2 (COVID-19) prevention and protection. The ultimate goal is to design prospective larger behavioral studies (SuRe first or R21) with a multi-centered intervention with other RTRN institutions to demonstrate the applicability of this approach specifically focusing on the AA/POC community.

DETAILED DESCRIPTION:
Several studies have shown that COVID-19 patients with co-existing diabetes were more likely to develop severe or critical disease conditions with more complications, and had higher incidence rates of antibiotic therapy, non-invasive and invasive mechanical ventilation, and death. Another important finding is that African Americans (AA)/People of Color (POC) are disproportionately impacted by COVID-19 to an extent not observed in other racial/ethnic subgroups. Diabetes Self-Management Education and Support (DSMS/S) facilitates the knowledge, skills, and ability necessary for diabetes self-care as well as activities that assist a person in implementing and sustaining the behaviors needed to manage their condition on an ongoing basis. Now, given the implications of COVID-19 on the AA/POC diabetes community, it is imperative to enhance DSME/S with education about protection and prevention of COVID-19. We will adapt and implement the "emPOWERed to Change" DSME/S program to provide enhanced type 2 diabetes mellitus (T2DM) education with an additional emphasis on COVID-19 protection and prevention. The proposed hypothesis, based on the Health Belief Model (HBM) and the Theory of Planned Behavior (TPB), is: African Americans (AA)/People of Color (POC) in Los Angeles County with type 2 diabetes mellitus (T2DM) randomized to participate in the "emPOWERed to Change" program (N=48) are more likely to demonstrate sustained glycemic control, increase in knowledge and skills related behaviors, and risk factors associated with T2DM and SARS-CoV-2 (COVID-19) and increased compliance with prevention, and vaccination as compared to those who are randomized to usual care (N=48) in this 12 week program.

Aim 1: to determine the efficacy of the "emPOWERed to Change" program on the knowledge and skills related to eating habits, physical activity, stress management, and medication adherence in the AA/POC population with type 2 diabetes.

Hypothesis: we hypothesized that AA/POC participants randomized to the program will have 20% increased knowledge and skills related to eating habits, physical activity, stress management, medication adherence, and control of diabetes compared to those randomized to the usual care.

Aim 2 to determine the effect of the "emPOWERed to Change" program on the knowledge related to T2DM and COVID-19 (risk factors, prevention of infection, COVID-19 vaccines, and access resources for vaccination) and compliance with prevention and vaccination against COVID-19.

Hypothesis: we hypothesized that AA/POC participants randomized to the program will have 20% increase in knowledge related to T2DM and COVID-19, compliance with prevention and vaccination against COVID-19 compared to those randomized to the usual care.

We propose a randomized control study design among 96 participants with 48 assigned to an intervention group and 48 assigned to a control group. This study will also explore the experience of the participants' appraisal of knowledge and skills acquisition for DSME/S to maintain T2DM control, reduce complications, and SARS-CoV-2 (COVID-19) prevention and protection. The ultimate goal is to design prospective larger behavioral studies (SuRe first or R21) with a multi-centered intervention with other RTRN institutions to demonstrate the applicability of this approach specifically focusing on the AA/POC community.

The presence of diabetes mellitus, hypertension, and obesity significantly increases the risk for hospitalization and death in COVID-19 patients. COVID-19 patients with diabetes were found to be more likely to develop severe or critical disease conditions with more complications and had higher incidence rates of antibiotic therapy, non-invasive and invasive mechanical ventilation, and death (Zhang, et al., 2020). In light of these findings, the potential that existing racial and ethnic disparities will be worsened and compounded by COVID-19 because African Americans continue to suffer a disproportionate burden of chronic diseases, with more pronounced disparities in type 2 diabetes, congestive heart failure, and hypertension.

Health disparities among AAs has continued and have shown to be perpetuated by the COVID-19 pandemic. California's death rate among African Americans is disproportionate as compared to representation in the population (10% mortality versus 6% population) and even more disproportionate in some counties. Specifically, the data from Los Angeles County showed a 14% mortality rate among African Americans, who make up 9% of the county's population (Azar, et al., 2020). In the context of circumstances surrounding COVID-19, the California Health Care Foundation identifies this pandemic as "a perfect storm of irrefutable evidence that people of color are caught in a web of social inequality." (Hernández, 2020) DSME/S is a crucial element in helping patients navigate and incorporate successful care into their daily lives. It has been proven to: instill lifestyle modifications which are directly associated with improved blood sugar control, reduce risk of diabetes complications, fewer hospitalizations, lower diabetes related medical cost and to be cost-effective. Some reports show that less than 38% of patients diagnosed with diabetes actually receive DSME/S (Torres, Tiwari, Movsas, Carrasquillo & Zonszein, 2015). The proposed study and intervention seek to consider and begin to mitigate these confounding issues.

As the COVID-19 pandemic appears to be ending among some populations, research suggests that AAs continue to be severely impacted. In communities that have higher percentages of AAs, study findings indicate an association between negative COVID-19 health outcomes and AAs, including higher prevalence and higher death rates. In addition, the data suggests that the odds of surviving the epidemic may correlate to poverty levels, indicating that other at-risk minority populations, affected by poverty, may also be disproportionately affected (Cyrus et al., 2020). Snowden and Graaf (2021) report that there are greater African American COVID-induced challenges and suffering, and COVID-19 threatens to perpetuate these differences.

While it is understood that policies are fundamental to shifting the trajectory of the Diabetes epidemic and the COVID-19 pandemic, we believe that COVID-19 education enhanced DSME/S interventions are promising. Moreover, we believe that by incorporating community-based outreach, testing, and access to culturally competent educational interventions within African American communities hold great promise for increased protection and prevention against COVID-19 along with better T2DM outcomes. This will in turn have a positive impact on some of the observed disparities. This research project can provide the groundwork to further develop and implement DSME/S that is easily accessible and less limiting than traditional DSME/S programs for this population, especially during a critical inflection point in the COVID-19 pandemic.

Literature suggests digital technology is the next link to enhanced communication between providers and patients. Patients with diabetes often report a variety of barriers to accessing DSME/S, especially issues with transportation and time commitments in attending on-site DSME/S programs. This online T2DM education program provides an alternative for those who are unable or unwilling to attend traditional DSME/S. While an online program does not replace the need for traditional DSME/S or certified diabetes educators, having online/on-demand availability does provide an additional resource for providers to offer for educating patients with diabetes in self-management and COVID-19 prevention and protection education.

The "emPOWERed to Change" program presents a unique, novel and timely approach to DSME/S with the enhancement of COVID-19 education. The program leverages digital technology to better support patients. It will be delivered virtually, on-demand, with culturally sensitive content and utilize mHealth and social media which has shown to be increasingly useful given the COVID-19 pandemic while capitalizing on the current trends of preferred engagement via technology for this population.

The "emPOWERed to change program" also integrates support through the use of Social media. This interaction provides an additional means for assisting patients with diabetes as it increases access to care, provides tools for self-management, and fosters support from others diagnosed with the same disease (Kenny, 2014). According to Power and Pitfalls of Social Media in Diabetes Care, (McMahon, 2013) some individuals find extra value in interacting with their peers online, as they may feel their provider lacks the ability to relate to them in the way other patients with diabetes can. Providers report finding that when patients utilize social media for support, they have become increasingly compliant with treatment recommendations, and appear to sustain healthy lifestyle changes (Cooper & Kar, 2014). These lifestyle changes include healthy eating and engaging in physical activity more often when these individuals have the support of their peers, and these peers, in many cases, are available exclusively online (Cooper & Kar, 2014). Also, engagement of individuals with diabetes via social media has been shown to provide the foundation for patients modified treatment regimens (McMahon, 2013).

While behavior modification plays an important role in controlling blood sugars, the use of technology can support self-management techniques and behaviors helpful to patients self-monitoring their blood glucose levels (Park, Burford, Nolan, & Hanlen, 2016).

Preliminary data from The Suga Project Foundation's DSME/S program, led by Natalie Pauls, PI, has shown that the elements of the "emPOWERed to Change" program are effective at increasing knowledge about type 2 diabetes, helping avoid risks of complication, improved communication with healthcare providers and an overall increased sense of better well-being through stress management and peer support.

Literature reviews by Cotter, et al., (2014) and Gabarron, et al., (2018) suggests that technology-enabled strategies provide a viable option for facilitating diabetes self-management, however, future research is needed on the use of web-based interventions in underserved communities, which is what this study will attempt to begin examining.

Study Design We propose a randomized, controlled study design among 134 participants. Through a simple randomization methodology, half of participants will be randomized to an intervention program and usual care group. The proposed hypothesis, based on the Health Belief Model (HBM) and the Theory of Planned Behavior (TPB), is: African Americans (AA)/People of Color (POC) in Los Angeles County with type 2 diabetes mellitus (T2DM) who participate in the "emPOWERed to Change" program will demonstrate sustained glycemic control.

(HbA1c<7%) and increase in knowledge of the risk factors associated with T2DM and SARS-CoV-2 (COVID-19) and increased adherence to medication and compliance with prevention, and vaccination as compared to those in the usual care group.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older African American, Male or Female, must be diagnosed with type 2 diabetes mellitus and be from MLK-OPC, no prior formal DSME/S program participation and must have internet access

Exclusion Criteria:

* Under 18 years of age, POC but not African American, not diagnosed with type 2 diabetes mellitus, not a patient of LAC DHS MLK-OPC facilities, not having internet access, had or receiving formal DSME/S program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-10 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Type 2 Glycemic Control - HbA1c of 7% or less | 12 weeks
  Achieve Glycemic control defined as an HbA1c of 7% or less

SECONDARY OUTCOMES:
Understanding of Diabetes Self-Management | 12 weeks
  Exhibit increased knowledge and skills as it relates to eating habits, physical activity, stress management, and medication adherence as measured by the DSMQ
Understand of COVID-19 Risks, Protection and Prevention | 12 weeks
  Exhibit increased knowledge related to risk factors associated with T2DM and COVID-19, prevention of infection, available resources and COVID-19 vaccines, and access resources for vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Jay Vadgama, M.D., Principal Investigator — Charles Drew University of Medicine and Science

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abazari P, Vanaki Z, Mohammadi E, Amini M. Inadequate investment on management of diabetes education. J Res Med Sci. 2012 Aug;17(8):792-8. PMID 23798949
- [Background] Azar KMJ, Shen Z, Romanelli RJ, Lockhart SH, Smits K, Robinson S, Brown S, Pressman AR. Disparities In Outcomes Among COVID-19 Patients In A Large Health Care System In California. Health Aff (Millwood). 2020 Jul;39(7):1253-1262. doi: 10.1377/hlthaff.2020.00598. Epub 2020 May 21. PMID 32437224
- [Background] Cooper, A., & Kar, P. (2014). A new dawn: The role of social media in diabetes education. Journal of Diabetes Nursing, 18(2), 68-71
- [Background] Cyrus E, Clarke R, Hadley D, Bursac Z, Trepka MJ, Devieux JG, Bagci U, Furr-Holden D, Coudray M, Mariano Y, Kiplagat S, Noel I, Ravelo G, Paley M, Wagner EF. The Impact of COVID-19 on African American Communities in the United States. Health Equity. 2020 Oct 30;4(1):476-483. doi: 10.1089/heq.2020.0030. eCollection 2020. PMID 33269331
- [Background] Gabarron E, Arsand E, Wynn R. Social Media Use in Interventions for Diabetes: Rapid Evidence-Based Review. J Med Internet Res. 2018 Aug 10;20(8):e10303. doi: 10.2196/10303. PMID 30097421
- [Background] Hernández SR , C. K . COVID-19: a perfect storm of health care inequality. Oakland (CA): California Health Care Foundation; 2020 Apr 10 [cited 2021 May 31]. From: https://www.chcf.org/blog/covid-19-perfect-storm-health-care-inequality/
- [Background] Kenny, C. (2014). Information technology, education and diabetes. Diabetes & Primary Care, 16(3), p. 111-112.
- [Background] Kitsiou S, Pare G, Jaana M, Gerber B. Effectiveness of mHealth interventions for patients with diabetes: An overview of systematic reviews. PLoS One. 2017 Mar 1;12(3):e0173160. doi: 10.1371/journal.pone.0173160. eCollection 2017. PMID 28249025
- [Background] Los Angeles County Department of Public Health. COVID-19 racial, ethnic, and socioeconomic data and strategies report [Internet]. Los Angeles (CA): LA County Department of Public Health; 2020 Apr 28 [cited 2021 May 31]. http://www.lapublichealth.org/docs/RacialEthnicSocioeconomicDataCOVID19.pdf
- [Background] McMahon, K. L. (2013). Power and Pitfalls of Social Media in Diabetes Care. Diabetes Spectrum, 26(4), 232-235. doi:10.2337/diaspect.26.4.232
- [Background] Park S, Burford S, Nolan C, Hanlen L. The Role of Digital Engagement in the Self-Management of Type 2 Diabetes. Health Commun. 2016 Dec;31(12):1557-65. doi: 10.1080/10410236.2015.1089468. Epub 2016 Apr 28. PMID 27124817
- [Background] Public Policy Institute of California (2021). California's Digital Divide. https://www.ppic.org/publication/californias-digital-divide/
- [Background] Snowden LR, Graaf G. COVID-19, Social Determinants Past, Present, and Future, and African Americans' Health. J Racial Ethn Health Disparities. 2021 Feb;8(1):12-20. doi: 10.1007/s40615-020-00923-3. Epub 2020 Nov 23. PMID 33230737
- [Background] Torres, E. A., Tiwari, A., Movsas, S., Carrasquillo, I., & Zonszein, J. (2015). Underutilization of Diabetes Education. Experience in an Urban Teaching Hospital in The Bronx. J Diabetes Metab Syndr Disord, 2(005).
- [Background] Zhang Y, Cui Y, Shen M, Zhang J, Liu B, Dai M, Chen L, Han D, Fan Y, Zeng Y, Li W, Lin F, Li S, Chen X, Pan P; medical team from Xiangya Hospital to support Hubei, China. Association of diabetes mellitus with disease severity and prognosis in COVID-19: A retrospective cohort study. Diabetes Res Clin Pract. 2020 Jul;165:108227. doi: 10.1016/j.diabres.2020.108227. Epub 2020 May 22. PMID 32446795